CLINICAL TRIAL: NCT05349591
Title: Cryopreserved Polyclonal Regulatory T Cell (cePolyTregs) Immunotherapy in Islet Transplantation
Brief Title: cePolyTregs in Islet Transplantation
Acronym: cePolyTregs
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to feasibility challenges and following mutual agreement by JDRF CCTN and the Principal Investigator for Statement of Work 4 (SOW4), the study conducted by Dr. James Shapiro has been withdrawn/terminated.
Sponsor: University of Alberta (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Juvenile Diabetes Research Foundation Canadian Clinical Trial Network (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00117578
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Diabetes type1
Keywords: Islet Transplantation; cePolytregs; Cryopreserved; Immunotherapy; Diabetes treatment; Immunosuppression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The Participants in this arm receive islet transplant only and no cePolyTregs.
- Treatment (Experimental): Participants will receive cePolyTregs (target 400-1600 million, with a minimal acceptable dose of 100 million) two weeks post islet transplant and will be followed for 1 year after cePolyTregs infusion to assess the safety and preliminary efficacy of cePolyTregs therapy.
  Interventions: Biological: cePolytreg

INTERVENTIONS:
Biological: cePolytreg — The treatment group will receive cePolyTregs 2 weeks after islet transplantation as immunotherapy to improve islet survival and reduce the need for immunosuppression drugs.
  Arms: Treatment

SUMMARY:
The transplant of the insulin-producing cell into the liver (Islet transplant) has been proven an effective and valuable treatment for type 1 diabetics patients with poor blood sugar. However, Islet transplant is currently limited by the number of pancreas organ donors and the need for lifelong medication requirements such as antirejection drugs. The investigators have learned that Regulatory T cells (Tregs), a small subset of a cluster of differentiation 4+ (CD4+) T cells, have emerged as the major contributor to self-tolerance by preventing the initiation of unwanted immune activation and by suppressing ongoing immune responses to limit bystander tissue destruction. It has been suggested that infusion of Tregs before extensive graft damage may improve long-term graft outcomes. In this trial, we propose to study Analogous cryopreserved PolyTregs (cePolyTregs). cePolyTregs is a product with the same in vivo functionality to that of the non-cryopreserved PolyTregs.

DETAILED DESCRIPTION:
Type-1 diabetes mellitus (T1DM) occurs due to a loss of insulin production caused by the destruction of the insulin producing cells located in the human pancreas. Patients living with T1DM experience substantial complications from uncontrolled blood sugar levels. Insulin administration is a life-saving treatment but fails to replicate the dynamic and responsive control provided by a person's own insulin producing cells. Insulin therapies can also increase the risk of severe episodes of low glucose, which significantly impacts quality of life in these patients. Additionally, these therapies fail to completely prevent long-term complications from this devastating disease.

The transplant of the insulin producing cell into the liver (Islet transplant) has been proven an effective and valuable treatment for those with poor blood sugar. However, Islet transplant is currently limited by the number of pancreas organ donors and the need for lifelong medication requirements such as antirejection drugs.

Tregs are a subset of CD4+ T cells that function to maintain immune system homeostasis and preserve tolerance to self-antigens. The function of Tregs in maintaining immune tolerance can be harnessed through Treg cell therapy for treating various immunological diseases. Tregs have the ability to migrate to sites of inflammation and have over 30 different immune regulatory mechanisms to respond to different inflammatory conditions. Treg effector function appears to work by bystander suppression, regulating local inflammatory responses through a combination of cell-cell contact and suppressive cytokine production. Finally, Tregs have been shown to play a critical role in tissue repair. The discovery of the transcription factor FOXP3 in 2003 represented a major advance in Treg characterization. FOXP3 is essential for Treg cell lineage specification and directly contributes to Treg function. However, FOXP3 is an intracellular protein that cannot be used to isolate Tregs for therapeutic uses. Thus, methods for the isolation of Tregs must rely on the use of cell surface markers. The discovery of the inverse relationship between CD127 and FOXP3 expression led to the use of the CD4+CD127lo/- CD25+ cell surface phenotype for high-yield selection of a highly pure human Tregs population that is highly suppressive in vitro, thus providing the best source of FOXP3+ Tregs for adoptive immunotherapy.

Cryoperserved PolyTregs (cePolyTregs) is a new cellular therapeutic for allogeneic or autologous applications that have been studied so far for the treatment of acute respiratory distress syndrome (ARDS) associated with SARS-CoV-2 infection. A previous analogous product, PolyTregs, prepared using a similar methodology and only differed in final formulation, is thought to perform similarly in vitro and in vivo. The clinical experience with cePolyTregs is still limited; however, the analogous PolyTregs has been extensively used as an both allogeneic and autologous product in various clinical conditions, including graft-versus host disease (GvHD), Type 1 Diabetes, kidney transplant, systemic lupus erythematosus (SLE), and pemphigus vulgaris (PV). These experiences with autologous PolyTregs provides valuable insights to cePolyTregs.

We have used the analogous PolyTregs product in a clinical trial in subjects receiving islet transplant (PolyTregs in Islet Transplant study). A total of 16 participants were screened for eligibility for the study at the University of Alberta within the period of March 2018 to March 2021. The participants were divided in two cohorts. Cohort 1 received islet transplant using Alemtuzumab induction therapy with Etanercept and Anakinra anti-inflammatory therapy. Cohort 2 received islet transplant using Anti-Thymocyte Globulin (ATG) induction therapy with Etanercept and Anakinra anti-inflammatory therapy. The treatment groups of both cohorts received PolyTregs infusion at 6 weeks and 2 weeks post islet transplantation for Cohort 1 and Cohort 2, respectively. All participants in both cohorts were maintained on low dose tacrolimus (Tac) and sirolimus (SRL) immunosuppression and were followed for a year after PolyTregs infusion to assess safety and preliminary efficacy of PolyTregs therapy. At the time of this protocol, 3 participants have received PolyTregs infusions. All reported AEs were mild to moderate in severity, resolved, and were determined to be unlikely or unrelated to PolyTregs infusion. While feasible, this trial was limited by the logistics issues surrounding PolyTregs manufacturing and the unpredictable nature of the timing of deceased donor islet transplant.

Cryopreserved PolyTregs (cePolyTregs) To facilitate feasibility surrounding logistics of PolyTregs manufacturing and the timing of islet transplant, cePolyTregs will be used. cePolyTregs is cryopreserved after its formulation and thawed immediately prior to infusion. cePolyTregs has a different formulation but the identity and characteristics are analogous to PolyTregs before and after cryopreservation. cePolyTregs will be delivered to the infusion site under controlled condition using a qualified shipper and will be kept cryopreserved until just prior to infusion. cePolyTregs will be first thawed in a water bath maintained at 34ºC - 38 ºC and kept on ice before administration. The thawed cePolyTregs product will be administered via a peripheral intravenous (IV) line primed with saline per established standard operating procedures. The product will be administered by peripheral IV line via manual syringe push in approximately 10 minutes to 30 minutes depending on the volume.

Following administration of the thawed cePolyTregs product, product bag, tubing and peripheral IV line will be flushed with normal saline to ensure complete dose is infused. Emergency medical equipment (i.e., emergency trolley) will be available during the infusion in case the subject has an allergic response, severe hypotensive crisis, or any other reaction to the infusion. Vital signs (temperature, respiration rate, pulse, and blood pressure) will be taken before and after infusion, then every 15 minutes (+/- 3 minutes) for at least one hour and until these signs are satisfactory and stable. The intravenous line will be maintained after the infusion and the subject will be asked to remain in the clinical research unit for 24 hours. Vital signs will be monitored every hour (+/- 3 minutes) for the first four hours and every four hours (+/- 3 minutes) thereafter.

Based on existing pre-clinical and clinical findings, we hypothesize that cePolyTregs protect from both auto and allorejection of transplanted islets, thereby improving insulin independent durability and C-peptide function over time in adults with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, subjects must be 18-68 years old, and have had T1DM for more than 5 years, complicated by at least 1 of the following situations that persist despite intensive insulin management efforts:

  1. Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels < 3.0 mmol/L, indicated by, 1 or more episodes of severe hypoglycemia requiring third party assistance within 12 months, or a Clarke score ≥4, or HYPO score ≥1000, or lability index (LI) ≥400 or combined HYPO/LI >400/>300.
  2. Metabolic instability, characterized by erratic blood glucose levels that interfere with daily activities and or 1 or more hospital visits for diabetic ketoacidosis over the last 12 months.

     In addition, participants must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

     Exclusion Criteria:
* Patients will be excluded if they meet any one or more of the following criteria:

  1. Severe co-existing cardiac disease, characterized by any one of these conditions: (a) recent myocardial infarction (within past 6 months); (b) left ventricular ejection fraction <30%; or (c) evidence of ischemia on functional cardiac exam
  2. Active alcohol or substance abuse (must be abstinent for 6 months prior to transplant)
  3. Clinical history of T1DM diagnosed >age 40, insulin dependent <5 years
  4. Active infection including Hepatitis C, Hepatitis B, HIV, TB (subjects with a positive PPD performed within one year of enrolment, and no history of adequate chemoprophylaxis)
  5. Measured glomerular filtration rate (GFR) < 60mL/min/1.73 m2
  6. Presence or history of macroalbuminuria (>300 mg/g creatinine)
  7. Clinical suspicion of nephritic (hematuria, active urinary sediment) or rapidly progressing renal impairment (e.g. Increase in serum creatinine of 25% within the last 3-6 months)
  8. Baseline Hb < 105g/L (<10.5 g/dL) in women, or < 120 g/L (<12 g/dL) in men
  9. Untreated proliferative retinopathy
  10. Positive pregnancy test, intent for future pregnancy, failure to follow effective contraceptive measures, or presently breast feeding
  11. Previous transplant or evidence of significant sensitization on PRA (at the discretion of the investigator).
  12. Insulin requirement >1.0 U/kg/day
  13. HbA1C >12%
  14. Uncontrolled hyperlipidemia [fasting LDL cholesterol > 3.4 mmol/L (133 mg/dL), treated or untreated; and/or fasting triglycerides > 2.3 mmol/L (90 mg/dL)]
  15. Under treatment for a medical condition requiring chronic use of steroids
  16. Use of coumadin or other anticoagulant therapy (except aspirin) or subject with PT INR > 1.5
  17. Untreated Celiac disease
  18. Patients with a Graves disease will be excluded unless previously adequately treated with radioiodine ablative therapy

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 58 weeks
  Any adverse event presented during the study

SECONDARY OUTCOMES:
Stimulated C-peptide level | Baseline
  Stimulated C-peptide response during Mixed Meal Tolerance Test (MMTT)
Stimulated C-peptide level | Day 30 post Islet transplantation
  Stimulated C-peptide response during Mixed Meal Tolerance Test (MMTT)
Stimulated C-peptide level | Day 90 post Islet transplantation
  Stimulated C-peptide response during Mixed Meal Tolerance Test (MMTT)
Stimulated C-peptide level | Week 58 post Islet transplantation
  Stimulated C-peptide response during Mixed Meal Tolerance Test (MMTT)

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD/PhD, Principal Investigator — University of Alberta; Indri Purwana, PhD, Study Director — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada